CLINICAL TRIAL: NCT02241590
Title: A Randomized, Placebo-Controlled, Double-Blind, Multi-Center Study to Assess the Efficacy and Safety of Fuzheng Huayu Combined With Entecavir in Liver Cirrhosis Patients Due to Hepatitis B Virus
Brief Title: Treatment of Liver Cirrhosis Due to Hepatitis B Virus With Fuzheng Huayu and Entecavir
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShuGuang Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Guangxi Ruikang Hospital (Other); Hubei Hospital of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); Huai'an No. 4 People's Hospital (Unknown); Ruijin Hospital (Other); Shenzhen Third People's Hospital (Other); Beijing Ditan Hospital (Other); Beijing YouAn Hospital (Other); China-Japan Friendship Hospital (Other); Tongji Hospital (Other); Wenzhou Central Hospital (Other); Jingmen No.1 People's Hospital (Other); Affiliated Hospital of Shandong Univercity of TCM (Unknown); The Ninth Hospital of Nanchang (Other); The People's Hospital of Ningxia (Other); Fifth Hospital of Shijiazhuang City (Other); The Fifth People's Hospital of Suzhou (Other); The Fifth People's Hospital of Anyang (Unknown)
Responsible Party: Principal Investigator, Liu Chenghai, Professor, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGHLC20140818001
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Liver Cirrhosis Due to Hepatitis B Virus
MeSH Terms: interventions — entecavir; fuzheng huayu

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entecavir + Placebo (Placebo Comparator): Tablet with Entrcavir+ Tablet with starch
  Interventions: Drug: Entecavir + Placebo
- Entecavir + Fuzheng Huayu Tablet (Experimental): Tablet with Entrcavir+ Tablet with Fuzheng Huayu
  Interventions: Drug: Entecavir + Fuzheng Huayu Tablet

INTERVENTIONS:
Drug: Entecavir + Placebo — The subjects will be taking 1 Entecavir tablet per day and 4 Placebo tablets three times a day for 48 weeks.
  Arms: Entecavir + Placebo
Drug: Entecavir + Fuzheng Huayu Tablet — The subjects will be taking 1 Entecavir tablet per day and 4 Fuzheng Huayu tablets three times a day for 48 weeks.
  Arms: Entecavir + Fuzheng Huayu Tablet

SUMMARY:
Liver Cirrhosis is a common pathological consequence of chronic liver disease. Hepatitis B Virus (HBV) is one of most etiologies of liver cirrhosis in China. The effective inhibition of HBV can partially stop or reverse liver fibrosis in patients with chronic Hepatitis and liver cirrhosis due to HBV, and the anti-fibrotic strategy focusing on the regulation of hepatic extracellular matrix is still required and hopefully improve the efficacy of anti-virals for liver fibrotic patients with HBV, especially is necessary for in the patients with advance fibrosis stage ie. liver cirrhosis. Fuzheng Huayu has been found to enhance the degradation of collagens in fibrotic liver and have a good action against liver fibrosis in patients with chronic hepatitis B. However, there are no high quality clinical evidences which can demonstrate if the combination of anti-viral and anti-fibrotic therapy can improve the reversion of liver cirrhosis due to HBV.

The primary objective of this study is to establish the safety and efficacy of the combination of Entecavir and Fuzheng Huayu for the reversion of liver fibrosis in patients with liver cirrhosis due to HBV.

ELIGIBILITY:
Inclusion Criteria:

* More than 6 months history of serum positive HBsAg
* Positive HBV-DNA
* Age 18-60
* Ishak fibrosis score of the biopsy within 6 months ≥5, no anti-virus or anti-fibrosis drug was taken within 6 months.
* Child-Pugh<7 (Stage A)
* The patient or the patient's guardian agrees to participate the trial and sign the informed Consent Form.

Exclusion Criteria:

* Primary Lamivudine, Adefovir dipivoxil and Entecavir resistance
* Decompensated liver cirrhosis
* HCC
* Liver histology conforming to other chronic liver diseases, such as moderate or severe non-alcoholic fatty liver disease(more than 1/3 steatosis in liver ), chronic hepatitis C, chronic hepatitis D, autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, inherited metabolic liver disease, drug or toxic induced liver injury, parasitic infections, alcoholic liver disease.
* Have psychiatric history or uncontrollable epilepsy patient.
* Uncontrollable diabetic patient
* History of hemoglobin disease (such as alpha- or beta-thalassemia, sickle cell disease, spherocytosis) or patients with toxic or autoimmune hemolytic anemia.
* Severe background disease like chronic respiratory failure, circulatory failure, kidney failure etc.
* In situ organ transplantation (such as liver, kidney, lung and heart) or bone marrow transplantation and stem cell transplantation.
* Immunocompromised patients: such as HIV infection or take immunosuppressor or glucocorticoid (such as cyclosporin, azathioprine, adrenocortical hormone) within 3 months or chemotherapy drugs (such as cyclophosphamide, ammonia and cancer chemotherapy) and radioactive therapy.
* Gestation or lactation period women and women who plan to get pregnant during the study period.
* Patient who are allergy to the experimental drug.
* Using history of anti-viral or anti-fibrosis drug within 6 months.
* Patients who are participating other trials.
* Other situation where PI thinks the patient should be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Degree of liver fibrosis | 48 weeks
  The collagen of liver tissue from 48 week post-treatment patients was stained. 3 pathologists read the slides independently and score the slides with Ishak system. If the Ishak score decrease 1 or more than 1 score, then it is recorded as regression.

CONTACTS AND LOCATIONS:
Overall Officials: Chenghai Liu, PhD, Study Director — ShuGuang Hospital
Locations (20):
- China (20):
  - Guangxi Ruikang Hospital, Nanning, Guangxi
  - The Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - The Fifth People's Hospital of Anyang, Anyang, Henan
  - Jingmen No.1 People's Hospital, Jingmen, Hubei
  - Hubei Hospital of TCM, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Hunan University of TCM, Changsha, Hunan
  - Huai'an No. 4 People's Hospital, Huai'an, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The Ninth Hospital of Nanchang, Nanchang, Jiangxi
  - Ningxia People's Hospital, Yinchuan, Ningxia
  - Affiliated Hospital of Shandong Univercity of TCM, Jinan, Shandong
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - Beijing Ditan Hospital Capital Medical University, Beijing
  - Beijing Youan Hospital Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - ShuGuang Hospital, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Shenzhen Third People's Hospital, Shenzhen

REFERENCES:
- [Derived] Li ZX, Zhao ZM, Liu P, Zheng QS, Liu CH. Treatment of HBV Cirrhosis with Fuzheng Huayu Tablet () and Entecavir: Design of a Randomized, Double-Blind, Parallel and Multicenter Clinical Trial. Chin J Integr Med. 2021 Jul;27(7):509-513. doi: 10.1007/s11655-020-3257-6. Epub 2020 Jun 22. PMID 32572776